CLINICAL TRIAL: NCT01765972
Title: Open Eye Corneal Swelling With Daily Disposable Contact Lenses and no Lens Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-5252
Record Dates: First submitted 2013-01-08; First posted 2013-01-11 (Estimated); Results first posted 2016-07-20 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2016-07

CONDITIONS: Corneal Swelling
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Test 1/Spectacles/Test 2/Test 3 (Other): Subjects assigned randomly to this arm will wear the study lenses sequentially as TEST 1 (etafilcon A with Lacreon), spectacles, TEST 2 (etafilcon A with Lacreon with print) and TEST 3 (etafilcon A with print) in both eyes for 8 +/-1 hours.
  Interventions: Device: etafilcon A with Lacreon; Device: etafilcon A with Lacreon with print; Device: etafilcon A with print; Device: Spectacles (habitual)
- Test 2/Test 3/ Spectacles/Test 1 (Other): Subjects assigned randomly to this arm will wear the study lenses sequentially as TEST 2 (etafilcon A with Lacreon with print), TEST 3 (etafilcon A with print), spectacles and TEST 1 (etafilcon A with Lacreon) in both eyes for 8 +/-1 hours.
  Interventions: Device: etafilcon A with Lacreon; Device: etafilcon A with Lacreon with print; Device: etafilcon A with print; Device: Spectacles (habitual)
- Test 3/Test 1/ Test 2/ Spectacles (Other): Subjects assigned randomly to this arm will wear the study lenses sequentially as TEST 3 (etafilcon A with print), TEST 1 (etafilcon A with Lacreon), TEST 2 (etafilcon A with Lacreon with print) and spectacles in both eyes for 8 +/-1 hours.
  Interventions: Device: etafilcon A with Lacreon; Device: etafilcon A with Lacreon with print; Device: etafilcon A with print; Device: Spectacles (habitual)
- Spectacles/Test 2/Test 1/Test 3 (Other): Subjects assigned randomly to this arm will wear the study lenses sequentially as spectacles, TEST 2 (etafilcon A with Lacreon with print), TEST 1 (etafilcon A with Lacreon) and TEST 3 (etafilcon A with print) in both eyes for 8 +/-1 hours.
  Interventions: Device: etafilcon A with Lacreon; Device: etafilcon A with Lacreon with print; Device: etafilcon A with print; Device: Spectacles (habitual)

INTERVENTIONS:
Device: etafilcon A with Lacreon — contact lens with Lacreon
  Other Names: Test 1
Device: etafilcon A with Lacreon with print — contact lens with Lacreon and cosmetic print
  Other Names: Test 2
Device: etafilcon A with print — contact lens with print
  Other Names: Test 3
Device: Spectacles (habitual) — Spectacles

SUMMARY:
The primary purpose of this clinical trial is to evaluate the eye's response to three test soft contact lenses as well as no lens wear, with respect to Corneal Staining.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. The subject must appear able and willing to adhere to the instructions set forth in the clinical protocol.
3. The subject must be between 18 and 45 years of age.
4. The subject must be an adapted soft contact lens wearer in both eyes.
5. The subject must be of East or Southeast Asian descent, e.g. ethnic Chinese, Japanese, Korean, Malay, Vietnamese, Indonesian, Filipino, etc. (it is preferred but not required that both the subject's biological parents are East or Southeast Asian ethnicity, by self report).
6. The subject's vertex corrected spherical equivalent distance refraction must be in the range of -1.00 to -6.00 D in each eye.
7. The subject's refractive cylinder must be no more than 1.00D in each eye.
8. The subject must have best corrected visual acuity of +0.14 logMAR (equivalent to 20/25-2) or better in each eye.
9. Subjects must own a wearable pair of spectacles and wear them on the day of the initial visit, during the washout before each phase and during the no lens wear phase.
10. The subject must have normal eyes (i.e., no ocular medications or infections of any type).

Exclusion Criteria:

1. Are currently pregnant or lactating by self report (subjects who become pregnant during the study will be discontinued).
2. Have any ocular or systemic allergies or diseases that may interfere with contact lens wear.
3. Have any systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but may not be limited to, diabetes. hyperthyroidism, recurrent herpes simplex/zoster, Sjogren's syndromes, xerophthalmia, acne rosacea, Stevens-Johnson syndromes, HIV/AIDS, hepatitis, and tuberculosis.
4. Use of any topical medications such aas eye drops or ointments.
5. Have entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosion, or aphakia.
6. Had any previous, or planned ocular or intraocular surgery (e.g. cataract surgery, radial keratotomy, PRK, LASIK, etc.).
7. Have any grade 2.0 or greater slit lamp findings (e.g. edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Efron classification scale or any other ocular abnormality that may contraindicate contact lens wear.
8. Have any known hypersensitivity or allergic reaction to one of the study products.
9. Have any ocular infection.
10. Have any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
11. Have participated in any contact lens or lens care product clinical trial within 14 days prior to study enrollment.
12. Have any infectious disease (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV by self report).
13. Currently wear their contact lenses on an extended wear basis.
14. Are an employee of the investigational clinic (e.g. Investigator, Coordinator, Technician)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 39 subjects were enrolled in this study. Of those enrolled subjects 15 subjects did not meet the eligibility criteria. The remaining 24 subjects were successfully dispensed a study lens and completed the study.
Groups:
- Test 1/Spectacle/Test 2/ Test 3: Subjects received Test 1 (etafilcon A with Laceron) and then received spectacle and then received Test 2 (etafilcon A with print) and then received Test 3 (etafilcon A with print).
- Test 2/ Test 3/ Spectacle/ Test 1: Subjects received Test 2 (etafilcon A with print) and then received Test 3 (etafilcon A with print) and then received spectacle and then received Test 1 (etafilcon A with Laceron).
- Test 3/ Test 1/ Test 2/ Spectacle: Subjects received Test 3 (etafilcon A with print) and then received Test 1 (etafilcon A with Laceron) and then received Test 2 (etafilcon A with print) and then received spectacle.
- Spectacle/ Test 2/ Test 1/ Test 3: Subjects received spectacle and then received Test 2 (etafilcon A with print) and then received Test 1 (etafilcon A with Laceron) and then received Test 3 (etafilcon A with print) .
Period: Overall Study
Arm/Group | Test 1/Spectacle/Test 2/ Test 3 | Test 2/ Test 3/ Spectacle/ Test 1 | Test 3/ Test 1/ Test 2/ Spectacle | Spectacle/ Test 2/ Test 1/ Test 3
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects that were dispensed a study lens.
Groups:
- Overall: All subjects that were dispensed a study lens.
Arm/Group | Overall
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.13 (2.437)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 24
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline of Corneal Swelling 8 Hours Post Fit
Description: Central corneal thickness was measured at baseline and 8-hour post fit with a modified optical pachometer on a Zeiss biomicroscope, interfaced to a PC. The pachometry measurement included seven readings; the computer is programmed to remove the high and low readings and to calculate the average of the remaining five readings. Only a single central corneal thickness measurement, the average of the 5 readings, was recorded by the investigator in the eCRF. The average percent change from baseline of corneal swelling was reported and was calculated as: ((Post fit - Baseline)/ Baseline) X 100.
Time Frame: 8 hours post fit
Population: Analysis population consists of subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Groups:
- Test 1 (Etafilcon A With Lacreon): Subjects that received Test 1 (etafilcon A with Lacreon) lens in any of the 4 periods of this study.
- Test 2 (Etafilcon A With Lacreon With Print): Subjects that received Test 2 (etafilcon A with Lacreon with print) lens in any of the 4 periods of this study.
- Test 3 (Etafilcon A With Print): Subjects that received Test 3 (etafilcon A with print) lens in any of the 4 periods of this study.
- Spectacle: Subjects that wore spectacles in any of the 4 periods of this study.
Arm/Group | Test 1 (Etafilcon A With Lacreon) | Test 2 (Etafilcon A With Lacreon With Print) | Test 3 (Etafilcon A With Print) | Spectacle
Number analyzed (Participants) | 24 | 24 | 24 | 24
percentage of change from baseline | 0.07 (0.288) | -0.02 (0.286) | 0.14 (0.350) | -0.06 (0.293)

ADVERSE EVENTS:
Time Frame: Entire duration of study (approximately 4 Months)
Groups:
- Spectacle: Subjects wore spectacles in any of the 4 periods of this study.
- Test 1 (Etafilcon A With Lacreon): Subjects received Test 1 (etafilcon A with Lacreon) in any of the 4 periods of this study.
- Test 2 (Etafilcon A With Lacreon With Print): Subjects received Test 2 (etafilcon A with Lacreon with print) in any of the 4 periods of this study.
- Test 3 (Etafilcon A With Print): Subjects received Test 3 (etafilcon A with print) in any of the 4 periods of this study.
Arm/Group | Spectacle | Test 1 (Etafilcon A With Lacreon) | Test 2 (Etafilcon A With Lacreon With Print) | Test 3 (Etafilcon A With Print)
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days